CLINICAL TRIAL: NCT03514017
Title: Phase II Trial of Ibrutinib and PD-1 Blockade in High Risk Chronic Lymphocytic Leukemia to Improve Immune Dysfunction
Brief Title: Ibrutinib and PD-1 Blockade in High Risk Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19199
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Results first posted 2023-09-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Lymphocytic; Leukemia; CLL; Blood disease; White blood cells; Bone marrow disease; Immunotherapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Hematologic Diseases; Bone Marrow Diseases | interventions — pembrolizumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Ibrutinib (Experimental): Treatment with pembrolizumab and ibrutinib and follow-up period of up to 24 months.
  Pembrolizumab is a humanized monoclonal antibody that blocks the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Ibrutinib is an inhibitor of Bruton's tyrosine kinase (BTK). Ibrutinib is a small-molecule inhibitor of BTK.
  Interventions: Drug: Pembrolizumab; Drug: Ibrutinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously (IV) at 200 mg every 3 weeks for 1 year and up to 2 years.
  Other Names: Keytruda®
Drug: Ibrutinib — Ibrutinib will be administered orally once daily at approximately the same time each day at the dose of 420 mg daily (3 capsules of 140 mg daily).
  Other Names: Imbruvica®

SUMMARY:
The purpose of this study is to evaluate the impact of sequential overlapping treatment with PD-1 monoclonal antibody (mAb), pembrolizumab/MK-1375, followed by ibrutinib on endogenous immune function in previously untreated, high-risk CLL patients. Immune function will be evaluated through various laboratory correlative tests.

ELIGIBILITY:
Inclusion Criteria:

* Have high risk CLL
* Have documented previously untreated CLL according to IWCLL criteria
* Willing and able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Demonstrate adequate organ function
* Able to take oral medication and willing to adhere to the medication regimen

Exclusion Criteria:

* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Meets IWCLL criteria to start therapy
* Has had any treatment for CLL including any investigational agent, chemotherapy, mAb, anti-PD-1, anti-PDL-1, or anti-CTLA-4
* Transformation of CLL to aggressive NHL (Richter's transformation or pro-lymphocytic leukemia)
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment
* Major surgery or a wound that has not fully healed within 4 weeks of first dose
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Chavez, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab and Ibrutinib: Treatment with pembrolizumab and ibrutinib and follow-up period of up to 24 months.
  Pembrolizumab is a humanized monoclonal antibody that blocks the interaction between PD-1 and its ligands, PD-L1 and PD-L2.
  Ibrutinib is an inhibitor of Bruton's tyrosine kinase (BTK). Ibrutinib is a small-molecule inhibitor of BTK.
  Pembrolizumab: Pembrolizumab will be administered intravenously (IV) at 200 mg every 3 weeks for 1 year and up to 2 years.
  Ibrutinib: Ibrutinib will be administered orally once daily at approximately the same time each day at the dose of 420 mg daily (3 capsules of 140 mg daily).
Period: Overall Study
Arm/Group | Pembrolizumab and Ibrutinib
Started | 5
Completed | 3
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Ibrutinib
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) to the Therapeutic Intervention
Description: Response categories according to The International Workshop on Chronic Lymphocytic Leukemia (IWCLL): Complete remission (CR); Complete remission with incomplete marrow recovery (CRi); Partial remission (PR); Progressive disease (PD); Stable disease (SD), defined as not meeting criteria for CR, CRi, PR or PD.
Time Frame: Up to 2 years
Population: evaluable participants
Measure: Number; unit: participants
Arm/Group | Pembrolizumab and Ibrutinib
Number analyzed (Participants) | 3
participants
  CR/PR | 2
  Stable Disease | 1

2. Primary Outcome: Time to Best Response
Description: Time to best response to chronic lymphocytic leukemia (CLL) to the therapeutic intervention.
Time Frame: Up to 2 years
Population: evaluable participants
Measure: Median (Standard Deviation); unit: months
Arm/Group | Pembrolizumab and Ibrutinib
Number analyzed (Participants) | 3
months | 3.02 (4.99)

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progressive disease (PD), defined as ≥ 50% rise in lymphocyte count to > 5 x10^9/L, ≥ 50% increase in lymphadenopathy, ≥ 50% increase in liver or spleen size, Richter's transformation, or new cytopenias due to CLL.
Time Frame: Up to 2 years
Population: Evaluable patients
Measure: Median (Standard Deviation); unit: months
Arm/Group | Pembrolizumab and Ibrutinib
Number analyzed (Participants) | 3
months | 16.57 (1.58)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of informed consent until 90 days after last dose of pembrolizumab and 30 days after last dose of ibrutinib, an average of 8.8 months. All-cause mortality was assessed through study completion, up to 24 months.
Arm/Group | Pembrolizumab and Ibrutinib
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Ibrutinib (N=5)
Gram negative sepsis (Infections and infestations) | 1 (1)
Aseptic Meningitis (Infections and infestations) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Ibrutinib (N=5)
Anemia (Blood and lymphatic system disorders) | 2 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (7)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (4)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (9)
Fever (General disorders) | 3 (5)
Chills (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (3)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (3)
Alanine aminotransferase increased (Investigations) | 4 (7)
Blood urea nitrogen increased (Investigations) | 1 (1)
Blood CO2 decreased (Investigations) | 1 (1)
Platelet count increased (Investigations) | 2 (2)
Neutrophil Count Increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (8)
Neutrophil count decreased (Investigations) | 2 (6)
Thyroid stimulating hormone increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Blood urea nitrogen decreased (Metabolism and nutrition disorders) | 1 (6)
Blood Urea Nitrogen Increased (Metabolism and nutrition disorders) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypochloremia (Metabolism and nutrition disorders) | 1 (2)
Iron decreased (Metabolism and nutrition disorders) | 1 (1)
Lactic Acid Increased (Metabolism and nutrition disorders) | 2 (2)
LDL increased (Metabolism and nutrition disorders) | 1 (1)
Serum protein decreased (Metabolism and nutrition disorders) | 2 (3)
Serm chloride decreased (Metabolism and nutrition disorders) | 2 (2)
Serum Chloride decreased (Metabolism and nutrition disorders) | 1 (1)
Total protein decreased (Metabolism and nutrition disorders) | 2 (4)
Uric acid decreased (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4)
Infections and Infestations -Other (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Macular wrinkle left eye (Eye disorders) | 1 (1)
Eye swelling/redness (Eye disorders) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Hypogammaglobulinemia (Immune system disorders) | 2 (3)
Squamous cell carcinoma, right calf (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nodule on dorsal aspect of left food (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03514017/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03514017/ICF_001.pdf